CLINICAL TRIAL: NCT03626233
Title: Study of the Physiology of Pre-eclampsia and Vascular Intrauterine Growth Restriction With Constitution of a Biological Collection
Brief Title: Study of the Physiology of Pre-eclampsia and Vascular IUGR With Constitution of a Biological Collection
Acronym: CPVP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: CPVP
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for maternal DNA sequencing and angiogenic factors (VEGF, PLGF, sFLt-1, sQDR) Urinary samples: Angiogenic factors Placenta: for placenta DNA sequencing and angiogenic factors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vascular group: Pregnant women with vascular pathology
  Interventions: Other: collect of placenta, blood and urinary samples at delivery
- Control group: * Pregnancy without any vascular complication
  * Delivery before or after 37 weeks of gestation (GW)
  * In case of delivery after 37GW: birth by cesarean delivery
  Interventions: Other: collect of placenta, blood and urinary samples at delivery

INTERVENTIONS:
Other: collect of placenta, blood and urinary samples at delivery — collect of placenta, blood and urinary samples at delivery

SUMMARY:
Preeclampsia and intrauterine growth retardation (IUGR) are serious and frequent pathologies, specific to pregnancy. They represent 70 000 new cases a year, or 9% of pregnancies and cause 50,000 premature births per year in France. The consequences in terms of morbidity and perinatal morbidity and the medical and economic costs make it an issue public health. Pre-eclampsia associates maternal hypertension with dysfunction kidney. There is no cure for pre-eclampsia or IUGR vascular during pregnancy. These pathologies invariably evolve towards a maternal and / or fetal aggravation sometimes very fast. Primary prevention and secondary education and screening for these pathologies are still insufficient. A better understanding of the pathophysiology of these placental vascular pathologies is necessary for the development of supported medical, obstetric and pediatric that will improve the state of health maternal and neonatal

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* With or without vascular pathology

Exclusion Criteria:

* refusal to participate
* multiple pregnancy
* major fetal malformation diagnosed during pregnancy follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: pregnant women with or without vascular pathology
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
genomic analysis on placenta | day of delivery
  by chromatin immunoprecipitation-sequencing (ChIP-seq)

SECONDARY OUTCOMES:
genomic analysis on blood | day of delivery
  by ChIP-seq
genomic analysis on placenta | day of delivery
  by immunohistochemistry an polymerase chain-reaction
VEGF blood level | day of delivery
PLGF blood level | day of delivery
sFlt1 blood level | day of delivery
sKDR blood level | day of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Lecarpentier, MD PhD, Principal Investigator — CHI CRETEIL
Locations (1):
- CHi Creteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No